CLINICAL TRIAL: NCT01922115
Title: The Effect of Anticholinergics on Cognitive Function in the Elderly: a Randomized Controlled Trial
Brief Title: The Effect of Anticholinergics on Cognitive Function in the Elderly
Acronym: ACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Urogynecologic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-1352
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Mental Competency; Urinary Bladder, Overactive; Cognitive Function
Keywords: COGNITIVE FUNCTION; OVERACTIVE BLADDER; [C23.888.942.343.780]
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TROSPIUM CHLORIDE (Active Comparator): Those with overactive bladder will be administered either a placebo or Sanctura XR extended release (Trospium chloride) for treatment (60 mg).
  Interventions: Drug: Trospium Chloride
- PLACEBO (Placebo Comparator): Subjects may be administered a placebo rather than the Sanctura XR (Trospium Chloride).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trospium Chloride — Subject will be administered either placebo or 60 mg dosage of Sanctura XR for treatment of overactive bladder. Subject will take Sanctura XR once every morning. Blood will be drawn for plasma extraction at each visit.
  Other Names: Sanctura XR
  Arms: TROSPIUM CHLORIDE
Drug: Placebo
  Arms: PLACEBO

SUMMARY:
Anticholinergic medication is used to treat overactive bladder (OAB). A known side effect of this medication is cognitive dysfunction. OAB is more prevalent in the elderly population - a group that also has a higher baseline risk of cognitive dysfunction. Our objective is to evaluate the effect of an anticholinergic medication on cognitive function in elderly women.

DETAILED DESCRIPTION:
Subjects will be randomized to: 1) trospium chloride or 2) placebo.

There are three aims:

1. To evaluate changes in cognitive function in elderly women taking trospium versus placebo, using validated cognitive assessment tests
2. To develop a useful battery of cognitive screening tests for monitoring the cognitive safety of OAB management
3. To understand how the timing of cognitive changes relates to the timing of improvement in OAB symptoms. The investigators will recruit 60 women aged ≥ 50 with the diagnosis of OAB. Cognitive assessments will be performed at baseline and Week 1 and 4 after drug initiation using paper-based validated questionnaires. OAB improvement will be assessed with validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female 50 or older
* Diagnosis of OAB (ICS definition)
* English literacy
* Ability to swallow oral medication
* Cognitive ability to give consent

Exclusion Criteria:

* Dementia/Depression/Delirium
* Current anticholinergic use (requires 2 week washout period)
* Current cholinesterase
* Urinary or gastric retention
* Severe decreased gastrointestinal motility
* Uncontrolled narrow-angle glaucoma
* Myasthenia gravis
* Diagnosis fo renal impairment (creatinine clearance <30 mL/min)

Ages: 50 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Geller, MD, Principal Investigator — UNC CHAPEL HILL
Locations (1):
- Unc Chapel Hill Urogynecology A2 Clinic, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Geller EJ, Dumond JB, Bowling JM, Khandelwal CM, Wu JM, Busby-Whitehead J, Kaufer DI. Effect of Trospium Chloride on Cognitive Function in Women Aged 50 and Older: A Randomized Trial. Female Pelvic Med Reconstr Surg. 2017 Mar/Apr;23(2):118-123. doi: 10.1097/SPV.0000000000000374. PMID 28067745

RESULTS

PARTICIPANT FLOW:
Groups:
- PLACEBO: Subjects may be administered a placebo rather than the Sanctura XR (Trospium Chloride).
  Placebo
Period: Overall Study
Arm/Group | TROSPIUM CHLORIDE | PLACEBO
Started | 28 | 31
Completed | 21 | 24
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TROSPIUM CHLORIDE | PLACEBO | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.39 (11.615) | 68.71 (10.615) | 68.56 (11.005)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 59
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7 | 25 | 32
  Black | 21 | 4 | 25
  Hispanic | 0 | 1 | 1
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hopkins Verbal Learning Test - Revised
Description: Assesses short term verbal learning and memory. Subscales include immediate recall (0-36) and delayed recall (0-12). Higher values indicate better outcomes.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TROSPIUM CHLORIDE | PLACEBO
Number analyzed (Participants) | 21 | 24
units on a scale
  Immediate Recall | 22.00 (5.51) | 24.38 (5.96)
  Delayed Recall | 6.71 (2.80) | 7.83 (3.28)

2. Secondary Outcome: Mini-Mental State Examination
Description: The mini-mental state examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia. The range is 0-30, with higher values indicating better outcomes.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TROSPIUM CHLORIDE | PLACEBO
Number analyzed (Participants) | 21 | 24
units on a scale | 28.14 (1.90) | 28.38 (1.76)

3. Secondary Outcome: Overactive Bladder Questionnaire
Description: The Overactive Bladder Questionnaire (OAB-q) was developed to assess symptom bother and the impact of overactive bladder (OAB) on health-related quality of life (HRQL). The instrument was developed and validated in both continent and incontinent OAB patients, including both men and women. Total range is 19-101 and higher values indicate worse outcomes.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TROSPIUM CHLORIDE | PLACEBO
Number analyzed (Participants) | 21 | 24
units on a scale | 41.45 (18.84) | 56.04 (20.21)

4. Primary Outcome: Hopkins Verbal Learning Test - Revised
Description: Assesses short term verbal learning and memory. See below for the subscale delayed recognition (0-24). Percentages of total responses correct are reported for delayed recognition, higher values indicate better outcomes.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: percentage of total correct
Arm/Group | TROSPIUM CHLORIDE | PLACEBO
Number analyzed (Participants) | 21 | 24
percentage of total correct | 81.68 (47.45) | 83.49 (26.72)

ADVERSE EVENTS:
Arm/Group | TROSPIUM CHLORIDE | PLACEBO
Serious Adverse Events (participants affected / at risk) | 2/28 | 0/31
Other Adverse Events (participants affected / at risk) | 10/28 | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TROSPIUM CHLORIDE (N=28) | PLACEBO (N=31)
Pulmonary Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blood Clot (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TROSPIUM CHLORIDE (N=28) | PLACEBO (N=31)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 4 (4) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry Eyes (Eye disorders) | 0 (0) | 1 (1)
Mood Swings (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No